CLINICAL TRIAL: NCT06189118
Title: Online Mindfulness-Based Cognitive Therapy vs Health Enhancement Program for Depressive Symptoms in Older Adults: a Randomized Controlled Trial
Brief Title: Online MBCT vs HEP for Depressive Symptoms in Older Adults: RCT
Acronym: OMH-D RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Professor, Geriatric Psychiatrist, Principal Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-884
Record Dates: First submitted 2023-09-11; First posted 2024-01-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Older Age; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Clinical Trial (n=100-120) older adults aged 60 and over who experience symptoms of depression (MADRS score 10 and more) and provide written consent will go through 1:1 stratified randomization (stratified cognition by Telephone-Montreal Cognitive Assessment, T-MoCA 19-25 and 26+points). The intervention will consist of 8 online sessions (90-min each) of Mindfulness based Cognitive Therapy. The active control will consist of 8 online sessions (90-min each) of Health Education Program. Participants in both study arms will continue with their usual antidepressant therapy and/or psychosocial care. Primary outcome: depressive symptoms; Secondary outcome: quality of life and cognition; Exploratory outcomes: anxiety and mindfulness presence. Baseline (weeks -2 to 0) and post-intervention (weeks 8-10) assessments will be conducted.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and outcome assessors will not be aware of allocation. Randomization and allocation will be conducted by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online Mindfulness based Cognitive Therapy (Experimental): The intervention will consist of 8 online weekly sessions (90-min each) of Mindfulness based Cognitive Therapy, plus daily home practice.
  Interventions: Behavioral: Online Mindfulness Based Cognitive Therapy or Health Education Program
- Online Health Education Program (Active Comparator): The active control will consist of 8 online weekly sessions (90-min each) of Health Education Program, plus daily home practice.
  Interventions: Behavioral: Online Mindfulness Based Cognitive Therapy or Health Education Program

INTERVENTIONS:
Behavioral: Online Mindfulness Based Cognitive Therapy or Health Education Program — 12 hours of online group training of Mindfulness Based Cognitive Therapy OR 12 hours of online group training of Health Education Program will be provided via teleconferencing. Additional both groups will perform daily home practice.
  Other Names: MBCT or HEP

SUMMARY:
In Canada, depression affects more than 300,000 adults over the age of 60, which costs the healthcare system an estimated $5 billion each year. Late-life depression (LLD) is associated with more deaths, more physical and mental health problems. LLD is hard to treat, as many people will not respond to treatment and many will stop taking antidepressant medication due to negative side-effects. Unfortunately, common non-medication treatments like cognitive behavioral therapy are often inaccessible because of long (6-12 months) wait times and high costs. In a previous study, we found that an 8-week group mindfulness-based cognitive therapy (MBCT) program improved depressive symptoms more than regular LLD treatment (i.e. antidepressants and/or support counseling). Now, a larger scale study is required to compare MBCT to an active control group. Furthermore, research and clinical experience during and post-Covid pandemic has shown that older adults are nowadays far less likely to participate in in-person intervention studies but appreciate and tolerate Zoom delivery of behavioral interventions. This study will compare the effects of MBCT versus an active control group, Health Enhancement Program (HEP), both delivered by Zoom, to see if it improves symptoms of depression in older adults. The study team plans to recruit approximately 100-120 participants in across Canada, who will be randomly assigned to 8-weeks of either MBCT or HEP, delivered by Zoom. The investigators will observe if these treatments improve depression as well as cognition by conducting in-person cognitive assessments. Currently there is a lack of affordable and accessible non-medication treatments for LLD that can be scaled to reach many people. If successful, Mindfulness may be a potential solution, as it is easily given in groups and is well-tolerated by older adults with LLD.

DETAILED DESCRIPTION:
Depression in older adults is associated with increased mortality, physical comorbidity, and neurocognitive decline. Up to 50-80% of patients are resistant to pharmacotherapy. Although psychotherapies such as cognitive behavioral therapy are effective for depression, such treatments are expensive and difficult to access, often with 6-12 month wait lists in Canada. There is a need for innovative non-pharmacological treatments for depression in older adults that are scalable and potentially cost-effective. Mindfulness-Based Cognitive Therapy (MBCT) stands out as a promising solution due to its scalable group format, good tolerability, and growing evidence of its efficacy in treating depression in adults. As well, clinical and research experience since Covid has shown that older adults have been much less likely to participate in in-person behavioral interventions.

Preliminary data in LLD: Our research group completed an 8-week intervention of MBCT (as an adjunct to treatment as usual =TAU) vs. TAU in older adults with depression +/- anxiety symptoms (N=61). MBCT was superior to TAU in improving depression scores (-7.9 (±4.4) vs. -4.0 (±4.7) point change, U = 179.5, p = 0.002), with a large effect size (d = 0.86). Furthermore, the investigators have conducted a number of pilot studies, which have established that older adults can feasibly use and enjoy behavioral interventions via teleconferencing. This study is the next step for a properly powered Phase III RCT (n=100-120) with an active comparator (HEP: Health Education Program) to establish the effectiveness of this novel intervention for LLD.

Research Aims:

Primary Objective: Using an 8-week RCT, assess whether MBCT improves scores of depressive symptoms scores compared to an active control (Health Enhancement Program (HEP)). Hypothesis 1A: The MBCT group will have a lower score in the Montgomery Asberg Depression Scale (MADRS) at 8-weeks, compared to HEP controls.

Secondary Objective: To investigate the effects of MBCT on cognitive function in older adults experiencing depression. Hypothesis 2A: MBCT will lead to higher scores in executive functioning and processing speed at 8 weeks. Hypothesis 2B: The MBCT group will have higher scores of quality of life (EQ-5D) scores at 8-weeks.

Exploratory Objective: To investigate effects of MBCT on scores of anxiety (GAD-7) and mindfulness presence (Five-Factor Mindfulness Questionnaire (FFMQ) Hypothesis 3A: The MBCT group will have reduced scores in the Generalized Anxiety Disorder 7 (GAD-7) at 8-weeks, compared to HEP controls. Hypothesis 3B: The MBCT group will have a higher score in mindfulness presence (FFMQ), compared to HEP controls.

Methods/Expertise: This study proposes an 8-week randomized controlled trial (RCT) for participants aged 60 years and older who score 10 or more points on the Montgomery Asberg Depression Scale (MADRS). An independent researcher will randomize participants, using computer software, stratified by baseline cognitive scores (T-MoCA: 19-25 and 26+ points), 1:1 to MBCT vs. an active control (HEP), virtually delivered via teleconferencing. This study will be a blinded to allocation (rater, investigator, and clinician) RCT. The investigators will conduct assessments of 1) depression scores (primary objective), 2) quality of life (EQ5D) cognition (neurocognitive battery), and 3) anxiety (GAD-7) and mindfulness (FFMQ) before and after virtually-delivered MBCT or HEP. Outcomes will be assessed at baseline and 8 weeks. The investigators have expertise in late-life mood disorders, mindfulness clinical trials, geriatric psychiatry, cognitive assessment, and biostatistics.

(all additional details can be found by section below)

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent (shown as to be able to explain back to the research assistant the purpose of the study as well as voluntary participation, rights, time commitments, etc.)
* MADRS score ≥ 10 (experiencing symptoms of moderate/severe depression) at baseline.
* Participants who have access to internet and basic digital skills to use their computer/tablet. -- Willing and able to attend ≥75% of MBCT or HEP sessions.
* Adequate understanding of English or French.
* Ability to sit for 90 minutes without discomfort.
* Willing to inform if any change is made to their psychotropic medications and dosage for the first 8 weeks of the study

Exclusion Criteria:

* cognitive deficits at baseline, as defined by T-MoCA score <19.
* diagnosis of post-traumatic stress disorder, bipolar I or II disorder, primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder), and/or severe personality disorder interfering with ability to function in a group setting intervention on a regular basis.
* substance abuse within the past 6 months.
* high suicide risk (e.g., active suicidal ideation and/or recent intent or plan).
* significant visual or hearing impairment
* significant impairments in fine motor skills.
* any medical illnesses that could prevent the participant from engaging in the intervention.
* history of psychiatric hospitalization in the last 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms scores | 8 weeks
  as measured by the Montgomery Asberg Depression Rating Scale

SECONDARY OUTCOMES:
Quality of Life scores | 8 weeks
  as measured by the EQ5D It is a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Processing Speed | 8 weeks
  as measured by the Trails Making Test A and WAIS-IV Digit Symbol (SDMT)
Executive Functioning | 8 weeks
  as measured by the trails Making Test B, WAIS- IV Digit Span and Verbal Fluency Test

OTHER OUTCOMES:
Exploratory outcomes: anxiety scores | 8 weeks
  Anxiety as measured by the Generalized Anxiety Disorder-7 scale
Exploratory outcome: Mindfulness Presence Scores | 8 weeks
  Mindfulness Presence as measured by the Five Facets of Mindfulness Questionnaire (FFMQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Mental Health University Institute, Verdun, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD available. Group, deidentified data may be requested directly to the PI by email.